CLINICAL TRIAL: NCT03228667
Title: QUILT-3.055: A Phase IIb, Multicohort, Open-Label Study of Combination Immunotherapies in Patients Who Have Previously Received Treatment With PD-1/PD-L1 Immune Checkpoint Inhibitors
Brief Title: QUILT-3.055: A Study of Combination Immunotherapies in Patients Who Have Previously Received Treatment With Immune Checkpoint Inhibitors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-803-02-17
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Urothelial Carcinoma; Head and Neck Squamous Cell Carcinoma; Merkel Cell Carcinoma; Melanoma; Renal Cell Carcinoma; Gastric Cancer; Cervical Cancer; Hepatocellular Carcinoma; Microsatellite Instability; Mismatch Repair Deficiency; Colorectal Cancer
Keywords: Pembrolizumab; Nivolumab; Non-Small Cell Lung Cancer (NSCLC); Immunotherapy; Interleukin-15; PD-1 Checkpoint Inhibitor; ALT-803; Atezolizumab; Avelumab; Small Cell Lung Cancer (SCLC); Urothelial Carcinoma; Head and Neck Squamous Cell Carcinoma (HNSCC); Merkel Cell Carcinoma (MCC); Melanoma; Renal Cell Carcinoma (RCC); Gastric Cancer; Cervical Cancer; Hepatocellular Carcinoma (HCC); Microsatellite Instability-High (MSI-H); PD-L1 Checkpoint Inhibitor; Mismatch Repair Deficient (dMMR) Solid Tumor Cancer; Colorectal Cancer (CRC); Durvalumab; PD-L1 t-haNK; N-803; Keytruda; Opdivo; Imfinzi; Bavencio; Tecentriq
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Transitional Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Merkel Cell; Melanoma; Carcinoma, Renal Cell; Stomach Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Microsatellite Instability; Turcot syndrome; Colorectal Neoplasms | interventions — ALT-803; pembrolizumab; Nivolumab; atezolizumab; avelumab; durvalumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Other): Patients with any of the cancers listed below who have progressed on or after single-agent checkpoint inhibitor therapy after experiencing an initial complete response (CR) or partial response (PR) while taking a checkpoint inhibitor.
  1a - Non-small cell lung cancer
  1b - Small cell lung cancer
  1c - Urothelial carcinoma
  1d - Head and neck squamous cell carcinoma
  1e - Merkel cell carcinoma
  1f - Melanoma
  1g - Renal cell carcinoma
  1h - Gastric cancer
  1i - Cervical cancer
  1j - Hepatocellular carcinoma
  1k - Microsatellite instability-high or mismatch repair deficient solid tumor cancer or colorectal cancer
  Interventions: Drug: N-803 + Pembrolizumab; Drug: N-803 + Nivolumab; Drug: N-803 + Atezolizumab; Drug: N-803 + Avelumab; Drug: N-803 + Durvalumab
- Cohort 2 (Other): Patients with NSCLC whose tumors have high PD-L1 expression (TPS ≥ 50%) and who relapsed on a PD-1 checkpoint inhibitor after experiencing an initial CR or PR when they received checkpoint inhibitor as a single-agent for first-line treatment.
  Interventions: Drug: N-803 + Pembrolizumab; Drug: N-803 + Nivolumab
- Cohort 3 (Other): Patients with NSCLC who had an initial CR or PR but subsequently relapsed on maintenance PD-1 checkpoint inhibitor therapy when they initially received checkpoint inhibitor therapy in combination with chemotherapy as first-line treatment.
  Interventions: Drug: N-803 + Pembrolizumab; Drug: N-803 + Nivolumab
- Cohort 4 (Experimental): Patients who are currently receiving PD-1/PD-L1 checkpoint inhibitor therapy and have disease progression after experiencing stable disease (SD) for at least 6 months during their previous treatment with PD-1/PD-L1 checkpoint inhibitor therapy.
  Interventions: Drug: N-803 + Pembrolizumab; Drug: N-803 + Nivolumab; Drug: N-803 + Atezolizumab; Drug: N-803 + Avelumab; Drug: N-803 + Durvalumab
- Cohort 5 (Experimental): Patients that have experienced disease progression by Investigator-assessment per irRECIST while receiving treatment in Cohorts 1-4.
  Interventions: Drug: N-803 + Pembrolizumab + PD-L1 t-haNK; Drug: N-803 + Nivolumab + PD-L1 t-haNK; Drug: N-803 + Atezolizumab + PD-L1 t-haNK; Drug: N-803 + Avelumab + PD-L1 t-haNK; Drug: N-803 + Durvalumab + PD-L1 t-haNK
- Cohort 6 (Experimental): Patients who have progressed after an initial response (CR or PR) to a PD-1/PD-L1 checkpoint inhibitor but now exhibit acquired resistance. They have received exactly one line of anti-PD-1 or anti-PD-L1 therapy (either pembrolizumab or nivolumab) for advanced NSCLC (Stage IV or recurrent).
  Interventions: Drug: N-803 + Docetaxel + Pembrolizumab; Drug: N-803 + Docetaxel + Nivolumab

INTERVENTIONS:
Drug: N-803 + Pembrolizumab — Patients will receive 200 mg pembrolizumab as an intravenous infusion over 30 minutes every three weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: N-803 + Nivolumab — Patients will receive 240 mg nivolumab as an intravenous infusion over 30 minutes every two weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: N-803 + Atezolizumab — Patients will receive 1200 mg atezolizumab as an intravenous infusion over 60 minutes every 3 weeks; if the first infusion is tolerated, subsequent infusions may be given over 30 minutes. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks.
  Arms: Cohort 1; Cohort 4
Drug: N-803 + Avelumab — Patients will receive 800 mg avelumab as an intravenous infusion over 60 minutes every 2 weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks.
  Arms: Cohort 1; Cohort 4
Drug: N-803 + Durvalumab — Patients will receive 10 mg/kg durvalumab as an intravenous infusion over 60 minutes every 2 weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks.
  Arms: Cohort 1; Cohort 4
Drug: N-803 + Pembrolizumab + PD-L1 t-haNK — Patients will receive 200 mg pembrolizumab as an intravenous infusion over 30 minutes every three weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks. Patients will receive PD-L1 t-haNK administered IV over 30 minutes at ~2 x 10^9 cells/dose weekly
  Arms: Cohort 5
Drug: N-803 + Nivolumab + PD-L1 t-haNK — Patients will receive 240 mg nivolumab as an intravenous infusion over 30 minutes every two weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks. Patients will receive PD-L1 t-haNK administered IV over 30 minutes at ~2 x 10^9 cells/dose weekly
  Arms: Cohort 5
Drug: N-803 + Atezolizumab + PD-L1 t-haNK — Patients will receive 1200 mg atezolizumab as an intravenous infusion over 60 minutes every 3 weeks; if the first infusion is tolerated, subsequent infusions may be given over 30 minutes. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks. Patients will receive PD-L1 t-haNK administered IV over 30 minutes at ~2 x 10^9 cells/dose weekly
  Arms: Cohort 5
Drug: N-803 + Avelumab + PD-L1 t-haNK — Patients will receive 800 mg avelumab as an intravenous infusion over 60 minutes every 2 weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks. Patients will receive PD-L1 t-haNK administered IV over 30 minutes at ~2 x 10^9 cells/dose weekly
  Arms: Cohort 5
Drug: N-803 + Durvalumab + PD-L1 t-haNK — Patients will receive 10 mg/kg durvalumab as an intravenous infusion over 60 minutes every 2 weeks. Patients will receive 15 µg/kg N-803 administered by subcutaneous injection every three weeks. Patients will receive PD-L1 t-haNK administered IV over 30 minutes at ~2 x 10^9 cells/dose weekly
  Arms: Cohort 5
Drug: N-803 + Docetaxel + Pembrolizumab — The study employs a 6-week cycle combination of: N-803 (1.2 mg flat dose SC), docetaxel (75 mg/m² IV - first 2 cycles only), and pembrolizumab (200 mg IV).
  Arms: Cohort 6
Drug: N-803 + Docetaxel + Nivolumab — The study employs a 6-week cycle combination of:N-803 (1.2 mg flat dose SC), docetaxel (75 mg/m² IV - first 2 cycles only), and nivolumab (240 mg IV). Nivolumab dosing may be increased to 480mg every four weeks as per the investigator's discretion.
  Arms: Cohort 6

SUMMARY:
QUILT-3.055 is a Phase 2b, open-label, multicohort study investigating combination immunotherapies in patients with advanced solid tumors who have previously been treated with PD-1/PD-L1 checkpoint inhibitors. The study aims to evaluate the safety and efficacy of NAI (nogapendekin alfa inbakicept) in combination with other agents like checkpoint inhibitors and cell therapies across various cancer types and treatment settings. The study includes multiple cohorts based on prior therapies and cancer types, with a focus on assessing overall response rate (ORR), overall survival (OS), and other measures of anti-tumor activity and immune response.

DETAILED DESCRIPTION:
All cohorts are closed to enrollment

ELIGIBILITY:
INCLUSION CRITERIA (Cohort 6 only)

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB/IEC guidelines.
3. Pathologically confirmed stage IV NSCLC disease.
4. Have received exactly 1 anti-PD-1 or anti-PD-L1 therapy (either pembrolizumab or nivolumab) for advanced disease (stage IV or recurrent disease, or stage I-III disease in certain circumstances) outlined below. Anti-PD-1 or anti-PD-L1 therapy may have been given alone or in combination with other therapy.

   a. For those participants who received neoadjuvant, adjuvant, and/or consolidation anti-PD-1 or anti-PD-L1 therapy for stage

   I-III disease:

   If they had disease progression within (≤) 365 days from initiation (cycle 1 day 1) of anti-PD-1 or anti-PD-L1 therapy, this counts as the single allowed anti-PD-1 or anti-PD-L1 therapy for advanced disease OR if they had disease progression more than (>) 365 days from initiation (cycle 1 day 1) of anti-PD-1 or anti-PD-L1 therapy, this is not considered anti-PD-1 or anti-PD-L1 therapy for advanced disease. These participants must have received anti-PD-1 or anti-PD-L1 therapy for stage IV or recurrent disease.
5. Have reported disease progression (in the opinion of the treating physician) more than (>) 84 days following initiation (cycle 1 day 1) of their most recent anti-PD-1 or anti-PD-L1 therapy (either pembrolizumab or nivolumab).
6. Participants who received anti-PD-1 or anti-PD-L1 therapy for stage IV or recurrent disease, must have had a best response of SD, PR or CR (in the opinion of the treating physician) on the anti- PD-1 or anti-PD-L1 therapy (either nivolumab or pembrolizumab) for stage IV or recurrent disease.
7. Participants with a known sensitizing mutation for which an - approved targeted therapy for NSCLC exists (e.g., EGFR, ALK, ROS1, BRAF, RET, NTRK, KRAS, HER2 and MET sensitizing mutations), must have previously received at least 1 of the approved therapy(s). Prior targeted therapy for participants with targetable alterations is allowed if all other eligibility criteria are also met.
8. ECOG performance status of 0 to 2.
9. Measurable tumor lesions according to RECIST v1.1.
10. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
11. Agreement to practice effective contraception for female participants of child-bearing potential and non-sterile males. Female participants of child-bearing potential must agree to use effective contraception for up 7 months after completion of therapy, and non-sterile male participants must agree to use a condom for up to 7 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), orals, injectables, 2 forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and hormonal therapy.

EXCLUSION CRITERIA (Cohort 6 only)

1. Systemic autoimmune disease currently requiring treatment (e.g., lupus erythematosus, rheumatoid arthritis, Addison's disease, or autoimmune disease associated with lymphoma). The participant must have been off treatment for 180 days.
2. History of organ transplant requiring immunosuppression; or history of pneumonitis or interstitial lung disease requiring treatment with systemic steroids; or a history of receiving systemic steroid therapy or any other immunosuppressive medication ≤ 3 days prior to study initiation. Daily steroid replacement therapy (eg, prednisone or hydrocortisone) and corticosteroids used to manage AEs are permitted.
3. History of known active hepatitis B or C infection.
4. Active infection requiring antibiotic therapy.
5. History of or active inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
6. Had major surgery within 28 days prior to study enrollment. Participants must have fully recovered from the effects of prior surgery in the opinion of the treating Investigator.
7. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute lymphocyte count < institutional ULN.
   2. Absolute neutrophil count (ANC) < 1,500 cells/mm3.
   3. Platelet count < 100,000 cells/mm3.
   4. Total bilirubin greater than the upper limit of normal (ULN; unless the participant has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or ALT (SGPT) > 1.5 × ULN.
   6. Alkaline phosphatase (ALP) levels > 2.5 × ULN.
   7. Hemoglobin < 9.0 g/dL.
   8. Serum creatinine > 2.0 mg/dL or 177 μmol/L or creatinine clearance < 40 mL/min (using the Cockcroft-Gault formula below): Female = [(140 - age in years) × weight in kg × 0.85] / [72 × serum creatinine in mg/dL] Male = [(140 - age in years) × weight in kg × 1.00] / [72 × serum creatinine in mg/dL]
8. Have any of following:

   1. Cirrhosis at a level of Child-Pugh B (or worse);
   2. Cirrhosis (any degree) and a history of hepatic encephalopathy; or
   3. Clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
9. Participation in an investigational drug study or history of receiving any investigational treatment within 30 days prior to the start of treatment on this study, except for hormone lowering therapy in participants with hormone-sensitive cancer.
10. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
11. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR, defined as Investigator-assessed CR + PR per RECIST v1.1. | Evaluated from the first dose of study drug and repeated at each scheduled disease-assessment visit for up to 24 months (or until progression/death), with the time-to-response summarized using Kaplan-Meier methods
  ORR reflects tumor shrinkage and is the key measure of antitumor activity.
Prolongation of OS with NAI therapy by ALC response, where: - OS is defined as the time from first study drug administration to death resulting from any cause. - ALC response is defined as achievement or maintenance of an on-treatment ALC ≥ 1,000 cells/μ | Measured from the date of the first study-drug administration to the date of death (any cause) and followed for up to 24 months after the last dose (or until death), allowing the correlation with on-treatment ALC changes
  OS is the gold-standard efficacy endpoint; the protocol explores whether an ALC rise predicts a survival benefit.

SECONDARY OUTCOMES:
ALC response to NAI therapy | From the date of first study-drug administration until the earlier of death or the planned end of follow-up, assessed up to 24 months.
  Defined as achieving a mean on-treatment absolute lymphocyte count (ALC) ≥ 1,000 cells/µL.
Prolongation of therapy | From the date of first study-drug administration until the earlier of death or the planned end of study follow-up, assessed up to 24 months after the last dose of study drug.
  Measured as the time on NAI treatment, analyzed according to whether the participant attained the ALC response described above.
Overall survival (OS) for all patients and subgroups | From the date of first study-drug administration until the earlier of death or the planned end of study follow-up, assessed up to 24 months after the last dose of study drug.
  Defined as the time from the first study-drug administration to death from any cause.
Disease-specific survival (DSS) | From the date of first study-drug administration until the earlier of death or the planned end of study follow-up, assessed up to 24 months after the last dose of study drug.
  Time from first study drug administration to death resulting from cancer.
Progression-free survival (PFS) | From the date of first study-drug administration until the earlier of death or the planned end of study follow-up, assessed up to 24 months after the last dose of study drug.
  Time from the first study-drug administration to either documented disease progression or death from any cause, whichever occurs first
Time to response | From the date of first study-drug administration until the earlier of death or the planned end of study follow-up, assessed up to 24 months after the last dose of study drug.
  The interval from the first dose of study drug to the first documented objective tumor response (CR or PR)
Duration of response (DoR) | From the date of first study-drug administration until the earlier of death or the planned end of study follow-up, assessed up to 24 months after the last dose of study drug.
  Time from the date of documented response (CR or PR) until disease progression or death.
Disease Control Rate (DCR): | Assessed at the end of each 6-week cycle (each cycle = 42 days) through 2 years (up to Cycle 17)
  measures the percentage of patients with stable disease (SD), partial response (PR), or complete response (CR). It indicates the proportion of patients who experience benefit from the treatment in terms of disease stabilization or tumor shrinkage.
Quality of life (QoL) - Assessed in cohorts 1-5 only. | From the date of first study-drug administration until the earlier of death or the planned end of study follow-up, assessed up to 24 months after the last dose of study drug.
  Assesses patient well-being using standardized questionnaires like EORTC QLQ-C30/LC13 or FACT PRO (module-specific), each with varying scales where higher scores generally indicate better functioning (but may also mean more symptoms).
Physical examinations | Baseline (screening), Day 1 (first dose), and prior to every subsequent NAI dose (e.g., every 2 weeks), then at each post-treatment safety visit (Week 12, Week 24, Week 36, Week 48, and at end-of-study visit)
  A full physical exam is conducted to assess any new or worsening clinical findings.

OTHER OUTCOMES:
Incidence of TEAEs and SAEs | Captured continuously from the first dose of study drug and monitored at every study visit throughout the treatment period and the post-treatment follow-up phase (until study closure, typically up to ~24 months after the last dose).
  All treatment-emergent adverse events and serious adverse events are recorded and graded using the NCI Common Terminology Criteria for Adverse Events version 5.0.
Laboratory tests | Baseline, Day 1, on-treatment (prior to each dose; every 2 weeks), and at each post-treatment safety visit (Week 12, Week 24, Week 36, Week 48, and end-of-study)
  Routine hematology, chemistry, and other safety-related labs are performed to detect treatment-related abnormalities.
Vital signs | Baseline, Day 1, before each NAI infusion (typically every 2 weeks), and at all scheduled safety follow-up visits (Week 12, Week 24, Week 36, Week 48, and final study visit)
  Blood pressure, heart rate, respiratory rate, temperature, and weight are recorded.
ORR (Objective Response Rate) | Assessed from the first dose onward at scheduled tumor-assessment visits (typically every 8-12 weeks) until progression, death, or study end (≈ 24 months).
  Cohorts 1-5 (irRECIST) Proportion of participants achieving a confirmed complete or partial response per immune-related RECIST.
PFS (Progression-Free Survival) | From Day 1 of first study-drug administration to first documented disease progression (per irRECIST/iRECIST) or death from any cause, whichever occurs first, assessed up to 24 months.
  Cohorts 1-5 (irRECIST) Time from first dose to disease progression (per irRECIST) or death from any cause, whichever occurs first.
Time to response | From Day 1 of first study-drug administration to the date of first confirmed complete or partial response, assessed up to 24 months.
  Cohorts 1-5 (irRECIST) Interval from first dose to the first documented objective response (CR or PR)
DCR (Disease-Control Rate) | Assessed at each tumor-assessment visit (baseline, Week 8 ± 1, Week 16 ± 2, Week 24 ± 2, and thereafter every 12 weeks) through 24 months.
  Cohorts 1-5 (irRECIST) Proportion of participants achieving CR, PR, or stable disease per irRECIST.
DoR (Duration of Response) | From the date of first confirmed response to subsequent disease progression or death, whichever occurs first, assessed up to 24 months.
  Cohorts 1-5 (irRECIST) Time from first documented response to disease progression or death.
Immunogenicity profile | Blood sampled at baseline, Day 1, Week 4, Week 12, and then every 12 weeks up to 24 months.
  Cohorts 1-5 (irRECIST) Detection of anti-drug antibodies or other immune responses to the investigational agents.
Cmax - Maximum plasma concentration of the investigational agent | Assessed on Cycle 1 Day 1 (each cycle = 28 days) and Cycle 2 Day 1. Sampling schedule on each study day: pre-dose, end-of-infusion, 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours, and 24 hours post-dose
  The highest observed plasma concentration of the study drug after a single intravenous infusion, expressed in ng · mL-¹. Concentrations are measured using a validated LC-MS/MS assay (lower limit of quantitation = 1 ng · mL-¹).
Tmax - Time to maximum plasma concentration of the investigational agent | Assessed on Cycle 1 Day 1 (each cycle = 28 days) and Cycle 2 Day 1. Sampling schedule on each study day: pre-dose, end-of-infusion, 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours, and 24 hours post-dose
  Time elapsed from the start of the infusion to the occurrence of Cmax, expressed in hours. Determined from the same plasma-sampling schedule used for Cmax.
AUC₀-t - Exposure (area under the plasma-concentration-time curve) from time 0 to the last quantifiable concentration | Assessed on Cycle 1 Day 1 (each cycle = 28 days) and Cycle 2 Day 1. Sampling schedule on each study day: pre-dose, end-of-infusion, 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours, and 24 hours post-dose
  Calculated using the linear-trapezoidal method applied to the concentration-time data obtained from the intensive sampling schedule (pre-dose through 24 h) on Cycle 1 Day 1. Units are ng · h · mL-¹.
AUC₀-τ - Steady-state exposure over one dosing interval | Assessed on Cycle 2 Day 1 (each cycle = 42 days). Intensive sampling: pre-dose, end-of-infusion, 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours post-dose. Sparse samples at weeks 12, 24, 36, 48, 60, 72, 84 (up to 24 months).
  Area under the plasma-concentration-time curve over a full dosing interval (τ) at steady state, calculated by the linear-trapezoidal method using pre-dose and post-dose samples collected on Cycle 2 Day 1 (or the first cycle where steady state is confirmed). Units: ng · h · mL-¹.
t½ - Terminal elimination half-life of the investigational agent | Determined from the same Cycle 1 Day 1 intensive sampling. No additional time points are required; the parameter is reported once per participant. The overall data-collection window for the participant is up to 24 months from first dose
  The time required for the plasma concentration to decline by 50 % during the terminal phase, calculated by log-linear regression of the last ≥3 measurable concentrations from the intensive sampling (typically 4 h, 8 h, 24 h) on Cycle 1 Day 1. Reported in hours.
ORR (Objective Response Rate) | Assessed from the first study-drug administration onward at scheduled tumor-assessment visits (typically every 8-12 weeks) and reported at the end of the follow-up period (up to the study's planned closure, e.g., ~24 months).
  Cohort 6 (iRECIST) Proportion of participants who achieve a confirmed complete response (CR) or partial response (PR) as assessed by the investigator using iRECIST criteria.
PFS (Progression-Free Survival) | From Day 1 of first study-drug administration to first documented disease progression (per irRECIST/iRECIST) or death from any cause, whichever occurs first, assessed up to 24 months.
  Cohort 6 (iRECIST) Time from the first dose of study drug to the first occurrence of disease progression (per iRECIST) or death from any cause, whichever comes first.
Time to response | From Day 1 of first study-drug administration to the date of first confirmed complete or partial response, assessed up to 24 months
  Cohort 6 (iRECIST) - Interval between the first study-drug administration and the date of the first documented objective response (CR or PR) per iRECIST.
DCR (Disease-Control Rate) | Assessed at each tumor-assessment visit (baseline, Week 8 ± 1, Week 16 ± 2, Week 24 ± 2, and thereafter every 12 weeks) through 24 months
  Cohort 6 (iRECIST) - Proportion of participants who achieve CR, PR, or stable disease (SD) according to iRECIST.
DoR (Duration of Response) | From the date of first confirmed response to subsequent disease progression or death, whichever occurs first, assessed up to 24 months.
  Cohort 6 (iRECIST) Time from the date of the first documented response (CR or PR) until disease progression (per iRECIST) or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Chan Soon-Shiong Institute for Medicine, El Segundo, California
  - MemorialCare Health System, Fountain Valley, California
  - Glendale Adventist Medical Center, Glendale, California
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Memorial Healthcare System, Hollywood, Florida
  - Miami Cancer Institute (Baptist Health South Florida), Miami, Florida
  - University of Miami, Miami, Florida
  - Horizon Oncology Associates, Lafayette, Indiana
  - University of Iowa Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Baptist Health - Lexington, Lexington, Kentucky
  - Baptist Health- Louisville, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota - Masonic Cancer Center, Minneapolis, Minnesota
  - Mercy Research Joplin, Joplin, Missouri
  - Mercy Clinic Cancer & Hematology - Chub O'Reilly Cancer Center, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Vincent Frontier Cancer Center (SCL), Billings, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic - Main Site, Cleveland, Ohio
  - Mercy Clinic Oklahoma City, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Gettysburg/Hanover Cancer Centers, Gettysburg, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Francis Cancer Center/Bon Secours St. Francis Health System, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Clinical Research, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Oncology Consultants of Houston, Houston, Texas
  - Bon Secours Richmond, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No